CLINICAL TRIAL: NCT03084484
Title: The Effect of Twice Daily Kiwifruit Consumption on Periodontal and Systemic Conditions Before and After Treatment: a Randomized Clinical Trial
Brief Title: Kiwifruit Effect on Periodontal Inflammation Kiwifruit Effect on Periodontal Inflammation
Acronym: PERIO-KIWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Filippo Graziani, DDS MClinDent PhD, Prof. of Periodontology, University of Pisa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 3729
Record Dates: First submitted 2017-03-03; First posted 2017-03-21 (Actual); Last update posted 2017-03-21 (Actual); Status verified 2017-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: Single-centre randomized, parallel design, clinical trial with a 5-month follow
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Subjects affected by periodontitis were examined and included in the study. After 2 months subjects also received non-surgical periodontal treatment and then followed for additional 3 months.
  Subjects in the test group were instructed to eat two kiwifruit per day during the whole study period.
  Interventions: Dietary Supplement: Kiwifruit addition to the diet; Procedure: Non Surgical periodontal treatment
- Control Group (Active Comparator): Subjects affected by periodontitis were examined and included in the study. After 2 months subjects also received non-surgical periodontal treatment and then followed for additional 3 months.
  Subjects in the control group didi not receive any dietary advice.
  Interventions: Procedure: Non Surgical periodontal treatment

INTERVENTIONS:
Dietary Supplement: Kiwifruit addition to the diet — Subjects were instructed to eat two kiwifruit per day during the whole study period. No recommendation on the type of kiwifruit, brand or origin was delivered. Kiwifruit was suggested to be taken as a whole and not mixed with sugar or other ingredients. No changes to their routinely dietary habits were suggested.
  Arms: Test Group
Procedure: Non Surgical periodontal treatment — Non-surgical treatment of periodontal pockets with hand and ultrasonic instrumentation

SUMMARY:
The importance of micronutrients has been extensively reviewed and it was concluded that for prevention and treatment of periodontitis daily nutrition should include sufficient antioxidants, vitamin D and calcium.

Up to now there is limited research available investigating the effect of vitamin C supplementation on the periodontal condition. Supplementation of vitamins and micronutrients has however raised numerous questions on clinical efficacy. Recently, a significant increase of medical literature on the effect of nutraceutical dietary aliments on general health has been noted.

the aim of the present study is twofold. The first objective is to investigate the effect of twice-daily kiwifruit consumption as sole treatment modality in untreated periodontitis, followed after two months by initial periodontal therapy supported by continued kiwifruit consumption. The second objective is to investigate the effect of twice daily kiwifruit consumption on periodontal and systemic parameters of these periodontitis patients 3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* proximal attachment loss of ≥3 mm in ≥2 non-adjacent teeth,
* PPD≥4 mm and bleeding on probing on at least 25 % of their total sites
* documented radiographic bone loss

Exclusion Criteria:

* younger than 18 years or older than 70 years,
* pregnant or lactating females,
* females using contraceptive pharmacological medications,
* reported diagnosis of any systemic illnesses including cardiovascular, renal, and liver diseases,
* in need of antibiotic treatment during initial periodontal treatment (IPT),
* IPT in the previous 6 months,
* allergic to latex, kiwifruit and fruits in general,
* suffering of eating or digestive disease or food intolerances,
* smoking more than 20 cigarettes per day.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Full-mouth bleeding score (FMBS) | Baseline, 2 months and 3 months after periodontal treatment
  Changes of FMBS. Unit of measure %

SECONDARY OUTCOMES:
Full-mouth plaque score (FMPS) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in FMPS. Unit of measure %
Pocket probing depth (PPD) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in PPD. Unit of measure: mm
Clinical attachment level (CAL) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in CAL. Unit of measure: mm
Recession of the gingival margin (REC) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in REC. Unit of measure: mm
Triglycerides | Baseline, 2 months and 3 months after periodontal treatment
  Changes in triglycerides. Unit of measure: mmol/L
Low-density lipoprotein (LDL) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in LDL. Unit of measure: mmol/L
High-density lipoprotein (HDL) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in HDL. Unit of measure: mmol/L
Cholesterol | Baseline, 2 months and 3 months after periodontal treatment
  Changes in total cholesterol, Unit of measure: mmol/L
Glycated Haemoglobin | Baseline, 2 months and 3 months after periodontal treatment
  Changes in Glycated haemoglobin. Unit of measure: mmol/mol
Vitamin C | Baseline, 2 months and 3 months after periodontal treatment
  Changes in Vitamin C. Unit of measure: µg/L
Systemic inflammation | Baseline, 2 months and 3 months after periodontal treatment
  Changes in C reactive protein (CRP). Unit of measure: mg/L
Systolic Blood Pressure (SBP) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in SBP Unit of measure: mmHg
Diastolic Blood Pressure (DBP) | Baseline, 2 months and 3 months after periodontal treatment
  Changes in DBP. Unit of measure: mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Filippo Graziani, Principal Investigator — filippo.graziani@med.unipi.it

REFERENCES:
- [Derived] Graziani F, Discepoli N, Gennai S, Karapetsa D, Nisi M, Bianchi L, Rosema NAM, Van der Velden U. The effect of twice daily kiwifruit consumption on periodontal and systemic conditions before and after treatment: A randomized clinical trial. J Periodontol. 2018 Mar;89(3):285-293. doi: 10.1002/JPER.17-0148. Epub 2018 Feb 27. PMID 29520772